CLINICAL TRIAL: NCT00588627
Title: Capsaicin Cough Sensitivity, Airway Inflammation and Neurogenic Peptides in Chronic Cough Associated With Postnasal Drip
Brief Title: Capsaicin Cough Threshold in Chronic Cough Due to Postnasal Drip
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Kaiser G. Lim, MD, Mayo Clinic
Other Study IDs: 2251-05; CR-20
Record Dates: First submitted 2007-12-25; First posted 2008-01-08 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Post Nasal Drip
Keywords: Chronic cough; Post nasal drip
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Mucus will be quantified and protease inhibitors will be added after collection. The specimen will be coded to deidentify. It will be transported to laboratory for storage and analysis. The mucus collected from the posterior nasopharynx will be frozen and assayed simultaneously. Substance P and Neurokinin A will be measured by ELISA at the end of the study period.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Post Nasal Drip and chronic cough
- 2: Post nasal drip and no cough

SUMMARY:
This study is being done to find out why some people with mucus dripping down the back of their throat have a nagging cough while others do not cough.

DETAILED DESCRIPTION:
The objective of the protocol is to determine the pathogenesis of cough in diseases of the aerodigestive tract. There were over 24 million ambulatory chronic cough visits nationally in 1991 and over 8,000 visits in 2004 at MCR. Current guidelines for chronic cough are based on case series and on empirical expert opinions. Studies have implicated mucosal inflammation, heightened sensitivity of capsaicin cough receptors on peripheral nerves and elaboration of inflammatory mediators including tussigenic neuropeptides. There are gaps in our knowledge of what triggers cough in many disease states. For example, postnasal drip syndrome has been estimated to account for 70% of chronic cough, yet it is known that not all patients with postnasal drip have chronic cough. Our hypothesis is that there must be critical factor/s that cause cough in one patient with postnasal drip but not in another. This study will evaluate whether there exists differences in capsaicin cough sensitivity, neuropeptides levels and mucosal inflammation in patients with postnasal drip and chronic cough and compared to its natural control group, subjects with postnasal drip with and without chronic cough. After standard therapy to eliminate postnasal drip, repeat measurement of capsaicin sensitivity and nitric oxide levels will be obtained. There is a critical need to determine the mechanisms underlying cough for better management. The study results will provide insight and fill gaps in our knowledge and will serve to advance future work evaluating mechanisms of cough in other disease states including asthma, GERD, interstitial lung disease and smokers.

ELIGIBILITY:
Inclusion Criteria:

-

Postnasal Drip with chronic cough:

1. Postnasal drip by rhinoscopy
2. Cough by visual analog scale.
3. Patients have to be 18 years old or older.
4. Cough-variant asthma must be excluded by a negative methacholine challenge test within one year, or documented failure of chronic cough to resolve after administration of inhaled corticosteroid (> one-month duration). Asthma is defined by the ATS guidelines.
5. Subjects must have a negative chest radiogram or Chest CT scan within 6 months.
6. No active GERD symptoms (< 7 RSI score) & a stable dose of Proton Pump Inhibitor (4 weeks).

   Eligibility Criteria of Postnasal Drip without cough:
7. Postnasal drip by rhinoscopy
8. No cough by visual analog scale.
9. Patients have to be 18 years old or older.

Exclusion Criteria:

* Subject Exclusion Criteria for Postnasal Drip with Chronic Cough:

  1. Presence of nasal polyposis and/or sinusitis or active GERD symptoms on examination.
  2. Current smokers (smoking within the 2 months prior to the study) will be excluded.
  3. Patients with an upper respiratory tract infection within the preceding 8 weeks.
  4. Patients taking angiotensin converting enzyme inhibitors.
  5. Patients on leukotriene receptor antagonist and/ or nasal topical corticosteroids or inhaled corticosteroids. Patient must be off nasal or inhaled corticosteroid by at least 4 weeks.

Exclusion Criteria: Same for Post Nasal Drip without cough except:

1. A chest radiogram is not necessary in this group.
2. Patients taking leukotriene inhibitors, or using nasal steroid therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic, community samples
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
We hypothesize that capsaicin cough sensitivity is increased in patients with PND-CC compared to subjects with PND without cough and that cough sensitivity to capsaicin will decrease with treatment for postnasal drip. | Endpoint

SECONDARY OUTCOMES:
We hypothesize that neurogenic inflammation is increased in patients with PND-CC compared to subjects with PND alone. | Endpoint
We hypothesize that nasal mucosal inflammation is increased in patients with PND-CC compared to subjects with PND alone, and that nasal mucosal inflammation will be decreased following treatment for postnasal treatment. | Endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Kaiser G. Lim, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States